CLINICAL TRIAL: NCT06807489
Title: Evaluation of the Risk of Developing Disordered Eating Behaviors or Eating Disorders in Children and Adolescents With Obesity Using a Digi-Physical Treatment Tool
Brief Title: Disordered Eating Risk in Pediatric Obesity Treatment Using a Digi-Physical Tool
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Evira AB (Industry)
Responsible Party: Principal Investigator, Pernilla Danielsson, Principal investigator, Karolinska Institutet
Other Study IDs: Evira200
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Childhood Obesity; Disordered Eating; Binge Eating Disorder; Anorexia Nervosa; Bulimia Nervosa
Keywords: Mobile Health; Support System; Self-Monitoring; Childhood Obesity; Childhood Obesity Treatment; Eating Disorder; Disordered Eating
MeSH Terms: conditions — Pediatric Obesity; Binge-Eating Disorder; Anorexia Nervosa; Bulimia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Digi-physical treatment group: Behavioral treatment combined with a digi-physical treatment tool for self- monitoring of weight and facilitating communication with the clinic. The patients are followed for three years from the start of treatment.
  Interventions: Device: Digi-physical treatment tool

INTERVENTIONS:
Device: Digi-physical treatment tool — A digital treatment tool named Evira will be used to provide the treatment.

SUMMARY:
The goal of this observational study is to evaluate the risk of developing disordered eating behavior or an eating disorder among children and adolescents with obesity who have used a digi-physical treatment tool with daily measurements conducted at home.

The primary outcomes are to:

* Evaluate the proportion of patients exhibiting documented signs of disordered eating behaviors during or after treatment (e.g., caloric restriction, skipping meals, binge eating).
* Evaluate the proportion of patients diagnosed with an eating disorder (e.g., anorexia nervosa, bulimia nervosa, binge eating disorder) during or after treatment.

Patients at Martina Childrens Hospital, Stockholm, Sweden, who have been treated with the digi-physical treatment tool will be included and their patient records will be reviewed for eating disorder diagnosis or a disturbed eating behavior.

DETAILED DESCRIPTION:
Children with chronic illnesses involving dietary restrictions as part of their treatment - such as obesity, diabetes mellitus, and celiac disease- are at an increased risk of developing eating disorders (ED) or disordered eating behaviors (DEB). Children with obesity are more likely to engage in unhealthy weight-control behaviors. Evidence-based, structured treatment programs for obesity do not elevate the risk of ED. On the contrary, such programs often intend to improve overall well-being. Professionally guided obesity treatment for children enhance self-esteem and has been shown to reduce both binge eating and loss of control over eating.

In this study, all participating children undergoing treatment for obesity will use a digi-physical treatment tool as a complement to behavioral treatment. This treatment tool includes daily measurements on a scale that does not show any digits, linked to a mobile app where weight development is shown as a moving average in the form of BMI standard deviation score (SDS). The app also provides an individualized target curve, visualizing the expected weight trajectory. Since weight changes in growing children are complex to interpret, BMI SDS is used as a standard metric. Objective data from the measuring device are automatically transferred to the database. Furthermore, direct communication between the clinic and the family is possible via the clinic interface and the app.

This study builds upon the investigators' previous one-year and three-year studies (ClinicalTrials.gov IDs: NCT04323215 and NCT06434259. The current follow-up study aims to evaluate the risk of developing DEB or an ED over a three-year period following the start of obesity treatment.

Approximately 400 children who have been treated with the digi-physical treatment tool will be included in the evaluation. Diagnoses and symptoms of DEB and ED will be retrieved from patient records.

ELIGIBILITY:
Inclusion Criteria:

* Obesity according to International Obesity Task Force (IOTF)
* Patients aged 6 years and older who have been treated with the digi-physical treatment tool

Exclusion Criteria:

* Patients with documented disordered eating behaviors or a diagnosed eating disorder prior to the start of treatment.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children aged 4-18 years who begin treatment for childhood obesity at Martina Children's Hospital in Stockholm, Sweden, and are treated with a digi-physical tool as a complement to behavioral therapy will be included. Only children with the possibility of receiving treatment for three years or more will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Disordered Eating Behaviors | From start of treatment to three years follow-up
  The proportion of patients exhibiting documented signs of disordered eating behaviors during or after treatment (e.g., caloric restriction, skipping meals, binge eating).
Referred patients | From start of treatment to three years follow-up
  The proportion of patients referred to another clinic for further evaluation of a potential eating disorder.
Diagnosis of Eating Disorder | From start of treatment to three years follow-up
  The proportion of patients diagnosed with an eating disorder (e.g., anorexia nervosa, bulimia nervosa, binge eating disorder).

SECONDARY OUTCOMES:
Time of Identification of Disordered Eating or Eating Disorder Diagnosis | From start of treatment to three years follow-up
  Identification of when, during the treatment process, signs of disordered eating or an eating disorder diagnosis are documented
Age of Onset of Eating Disorder | From start of treatment to three years follow-up
  The age at which the first documented signs of disordered eating behaviors or a diagnosed eating disorder occured.
Association with Neurodevelopmental Disorders | From start of treatment to three years follow-up
  Evaluation of the relationship between documented disordered eating behaviors or eating disorders and neurodevelopmental diagnoses, such as ADHD or autism.
Association with Mental Health Issues | From start of treatment to three years follow-up
  Examination of how documented signs of disordered eating behaviors or eating disorders are related to other mental health issues, such as stress, anxiety, or depression.
Change in BMI SDS During Treatment | From start of treatment to the last measurement, up to three-years
  Change in BMI SDS from the start of treatment as an indicator of treatment efficacy and its potential connection to disordered eating behaviors.
Measurement Frequency and Adherence | From start of treatment to three-years follow-up
  Analysis of how frequently patients perform the recommended daily measurements and how this correlates with the risk of disordered eating behaviors or other treatment outcomes.
Association with Curve Patterns | From start of treatment to the last measurement, up to three-years
  Analysis of the growth or weight curve patterns to identify potential factors indicating disordered eating behaviors or eating disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Pernilla Danielsson Liljeqvist, Associate Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Childrens Hospital Martina, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from Evira AB but restrictions apply to the availability of these data, which were used under license for the current study, and so are not publicly available. Data are however available from the authors upon reasonable request and with permission of Evira AB.

REFERENCES:
- [Background] Hagman E, Johansson L, Kollin C, Marcus E, Drangel A, Marcus L, Marcus C, Danielsson P. Effect of an interactive mobile health support system and daily weight measurements for pediatric obesity treatment, a 1-year pragmatical clinical trial. Int J Obes (Lond). 2022 Aug;46(8):1527-1533. doi: 10.1038/s41366-022-01146-8. Epub 2022 May 31. PMID 35641569